CLINICAL TRIAL: NCT01134861
Title: A Three-Arm Phase III Study of Concomitant Versus Sequential Chemotherapy and Thoracic Radiotherapy for Patients With Locally Advanced Inoperable Non-small Cell Lung Cancer
Brief Title: Radiation Therapy Plus Chemotherapy in Treating Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9410; U10CA021661 (NIH); CDR0000063640 (Other: Radiation Therapy Oncology Group)
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Etoposide; Vinblastine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Sequential ChemoRT (Active Comparator): Vinblastine 6 mg/m2 i.v. bolus weekly first 5 weeks Cisplatin 100 mg/m2 i.v. over 30-60 minutes, days 1 & 29 RT: 63 Gy/7 wks/34 daily fractions (1.8 Gy X 25 fx then 2.0 Gy X 9 fx) beginning day 50
  Interventions: Drug: cisplatin; Drug: Vinblastine; Radiation: Radiation therapy
- Arm 2: Concurrent STD RT (Experimental): Vinblastine 5 mg/m2 i.v. bolus weekly first 5 weeks Cisplatin 100 mg/m2 i.v. over 30-60 minutes, days 1 & 29 RT: 63 GY/7 wks/34 daily fractions (1.8 Gy X 25 fx then 2.0 Gy X 9 fx) beginning day 1
  Interventions: Drug: cisplatin; Drug: Vinblastine; Radiation: Radiation therapy
- Arm 3: Concurrent HFX RT (Experimental): Oral VP-16 50 mg b.i.d. X 10 only on RT treatment days 1-5, 8-12, 29-33, and 36-40 (76 mg/day if BSA < 1.7m2) Cisplatin 50 mg/m2 i.v. over 30-60 minutes on days 1, 8, 29, and 36 RT: 69.6 Gy/6 wks/58 X 1.2 Gy twice daily fractions (at least 6 hours apart) beginning day 1
  Interventions: Drug: Etoposide; Drug: Cisplatin; Radiation: Radiation therapy

INTERVENTIONS:
Drug: cisplatin — 100 mg/m2 i.v. over 30-60 minutes, days 1 & 29
  Arms: Arm 1: Sequential ChemoRT; Arm 2: Concurrent STD RT
Drug: Etoposide — Oral etoposide given 50 mg b.i.d. X 10 only on RT treatment days 1-5, 8-12, 29-33, and 36-40. 75 mg/day if body surface area < 1.7 m2
  Other Names: VP-16
  Arms: Arm 3: Concurrent HFX RT
Drug: Vinblastine — 5 mg/m2 i.v. bolus weekly first 5 weeks of RT
  Arms: Arm 1: Sequential ChemoRT; Arm 2: Concurrent STD RT
Radiation: Radiation therapy — 63 Gy/7 wks/34 daily fractions (1.8 Gy X 25 fx then 2.0 Gy X 9 fX) beginning day 50 of protocol treatment
  Arms: Arm 1: Sequential ChemoRT
Drug: Cisplatin — 50 mg/m2 i.v. over 30-60 minutes on days 1, 8, 29, and 36
  Arms: Arm 3: Concurrent HFX RT
Radiation: Radiation therapy — 63 Gy/7 wks/34 daily fractions (1.8 Gy X 25 fx then 2.0 Gy X 9 fx) beginning day 1 of protocol treatment
  Arms: Arm 2: Concurrent STD RT
Radiation: Radiation therapy — 69.6 Gy/6 wks/58 X 1.2 Gy twice daily fractions (at least 6 hours apart) beginning day 1 of protocol therapy
  Arms: Arm 3: Concurrent HFX RT

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of various schedules of radiation therapy and combination chemotherapy using vinblastine and cisplatin or cisplatin and etoposide in treating patients with stage II or stage III non-small cell lung cancer that cannot be removed surgically.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the survival rate of patients with locally advanced, unresectable non-small cell lung cancer randomized to concomitant vinblastine/cisplatin (VBL/CDDP) and thoracic radiotherapy versus sequential VBL/CDDP and once-daily thoracic radiotherapy. II. Compare the survival rate of such patients randomized to 2 courses of concomitant etoposide/cisplatin and hyperfractionated thoracic radiotherapy versus sequential VBL/CDDP and once-daily thoracic radiotherapy. III. Assess the frequency of treatment-related esophageal and hematologic toxicity/morbidity in patients on concomitant versus sequential chemoradiation treatment arms.

OUTLINE: Randomized study. The following acronyms are used: CDDP Cisplatin, NSC-119875 VBL Vinblastine, NSC-49842 VP-16 Etoposide, NSC-141540 Arm I: 2-Drug Combination Chemotherapy Followed by Radiotherapy. CDDP/VBL; followed by thoracic irradiation using photons of at least 6 MV (electrons may be used to boost the supraclavicular lymph nodes). Arm II: Radiotherapy plus 2-Drug Combination Chemotherapy. Thoracic irradiation using equipment as in Arm I; plus CDDP/VBL. Arm III: Hyperfractionated Radiotherapy plus 2-Drug Combination Chemotherapy. Thoracic irradiation using equipment as in Arm I; plus CDDP/VP-16.

PROJECTED ACCRUAL: A total of 597 patients will be entered over 3.1-4.2 years. If fewer than 6 patients/month are accrued, the feasibility of the study will be re-evaluated.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Locoregionally advanced, inoperable, non-small cell lung cancer with no evidence of distant metastases, i.e.: Stage II/IIIA medically inoperable disease Stage IIIA/IIIB unresectable disease No pleural effusion Appearance after an invasive thoracic procedure allowed No more than 5% weight loss within 3 months prior to diagnosis Confirmed N2 disease should first be evaluated for protocol RTOG-9309

PATIENT CHARACTERISTICS: Age: At least 18 Performance status: Karnofsky 70%-100% Hematopoietic: AGC at least 2,000 Platelets at least 100,000 Hemoglobin at least 8.0 g/dL Hepatic: (unless abnormality caused by benign disease) Bilirubin no more than 1.5 times normal AST no more than 1.5 times normal Renal: Creatinine no more than 1.5 mg/dL Cardiovascular: No myocardial infarction within the past 6 months No angina No congestive heart failure No uncontrolled arrhythmia Other: No synchronous or prior invasive malignancy within 3 years except nonmelanomatous skin cancer No pregnant women Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior thoracic or neck radiotherapy Surgery: No prior complete or nearly complete tumor resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 1994-07; Primary Completion 1998-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Overall Survival | from date of randomization to date of death or last follow-up for patients still alive

CONTACTS AND LOCATIONS:
Overall Officials: Walter J. Curran, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University

REFERENCES:
- [Background] Siddiqui F, Bae K, Langer CJ, Coyne JC, Gamerman V, Komaki R, Choy H, Curran WJ, Watkins-Bruner D, Movsas B. The influence of gender, race, and marital status on survival in lung cancer patients: analysis of Radiation Therapy Oncology Group trials. J Thorac Oncol. 2010 May;5(5):631-9. doi: 10.1097/jto.0b013e3181d5e46a. PMID 20432520
- [Background] Konski AA, Bhargavan M, Owen J, et al.: "Less is not always more": an economic analysis of Radiation Therapy Oncology Group 94-10. [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-1080, S182, 2007.
- [Background] Choy H, Swann S, Nabid A, et al.: Comparison of 5-year survival between RTOG-94-10 and a phase 2 study of induction chemotherapy followed by efaproxiral + radiotherapy in patients with locally advanced NSCLC. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-49, S28-9, 2006.
- [Background] Bradley J. A review of radiation dose escalation trials for non-small cell lung cancer within the Radiation Therapy Oncology Group. Semin Oncol. 2005 Apr;32(2 Suppl 3):S111-3. doi: 10.1053/j.seminoncol.2005.03.020. PMID 16015546
- [Background] Langer CJ, Swann S, Curran W, et al.: Reassessing prognostic factors in the era of combined modality therapy for locally advanced NSCLC: a retrospective analysis of RTOG 9410 and 9801. [Abstract] Int J Radiat Oncol Biol Phys 63 (2 Suppl 1): A-65, S39, 2005.
- [Background] Machtay M, Hsu C, Komaki R, Sause WT, Swann RS, Langer CJ, Byhardt RW, Curran WJ. Effect of overall treatment time on outcomes after concurrent chemoradiation for locally advanced non-small-cell lung carcinoma: analysis of the Radiation Therapy Oncology Group (RTOG) experience. Int J Radiat Oncol Biol Phys. 2005 Nov 1;63(3):667-71. doi: 10.1016/j.ijrobp.2005.03.037. Epub 2005 May 31. PMID 15927409
- [Background] Machtay M, Swann S, Komaki R, et al.: Overall treatment time during concurrent chemoradiotherapy and outcomes: an RTOG secondary analysis. [Abstract] Lung Cancer 50 (Suppl 2): A-O-042, S17, 2005.
- [Background] Machtay M, Swann S, Komaki R, et al.: What is the meaning of local-regional control after chemoradiation for locally advanced NSCLC? An RTOG analysis. [Abstract] Lung Cancer 50 (Suppl 2): A-O-041, S17, 2005.
- [Background] Swann RS, Machtay M, Komaki R, et al.: Impact of overall treatment time during concurrent chemoradiotherapy for locally advanced NSCLC: an RTOG secondary analysis. [Abstract] J Clin Oncol 23 (Suppl 16): A-7061, 635s, 2005.
- [Background] Werner-Wasik M, Scott C, Curran WJ, et al.: Correlation between acute esophagitis and late pneumonitis in patients (pts) with locally advanced non-small cell lung cancer (LA-NSCLC) receiving concurrent thoracic radiotherapy (RT) and chemotherapy: a multivariate analysis of the Radiation Therapy Oncology Group (RTOG) database. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1192, 2002.
- [Background] Sause W, Scott C, Byhardt R, et al.: Combined chemotheray radiation therapy treatment in unresected non-small cell lung cancer: Radiation Therapy Oncology Group (RTOG) experience. Lung Cancer 29(suppl 2): 2000.
- [Result] Curran WJ, Scott CB, Langer CJ, et al.: Long-term benefit is observed in a phase III comparison of sequential vs concurrent chemo-radiation for patients with unresected stage III nsclc: RTOG 9410. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2499, 2003.
- [Result] Langer CJ, Hsu C, Curran WJ, et al.: Elderly patients (pts) with locally advanced non-small cell lung cancer (LA-NSCLC) benefit from combined modality therapy: secondary analysis of Radiation Therapy Oncology Group (RTOG) 94-10. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1193, 2002.
- [Result] Langer CJ, Hsu C, Curran W, et al.: Do elderly patients (pts) with locally advanced non-small cell lung cancer (NSCLC) benefit from combined modality therapy? A secondary analysis of RTOG 94-10. [Abstract] Int J Radiat Oncol Biol Phys 51(3 suppl 1): A-36, 20-21, 2001.
- [Result] Movsas B, Scott C, Curran W, et al.: A quality-adjusted time without symptons or toxicity (QTWiST) analysis of Radiation Therapy Oncology Group (RTOG) 94-10. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1247, 313a, 2001.
- [Result] Curran WJ, Scott C, Langer C, et al.: Phase III comparison of sequential vs concurrent chemoradiation for patients with unresected stage III non-small cell lung cancer (NSCLC): initial report of Radiation Therapy Oncology Group (RTOG) 9410. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A1891, 2000.
- [Result] Komaki R, Seiferheld W, Curran W, et al.: Sequential vs. concurrent chemotherapy and radiation therapy for inoperable non-small cell lung cancer (NSCLC): analysis of failures in a phase III study (RTOG 9410). [Abstract] Int J Radiat Oncol Biol Phys 48 (3 suppl): A-5, 113, 2000.